CLINICAL TRIAL: NCT01883518
Title: Non-randomized Single-center Study Phase II Evaluating the Efficacy and Toxicity of Autologous Dendritic Cell Vaccine Loaded With Allogeneic Tumor Lysate Expression of Cancer Testis Antigens in Patients With Soft Tissue Sarcoma
Brief Title: Autologous Dendritic Cell Vaccine in Patients With Soft Tissue Sarcoma
Acronym: ADCVCTAST
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-01-2013
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Sarcoma; Neoplasms, Connective and Soft Tissue
Keywords: Fibrosarcoma; Neurofibrosarcoma; Histiocytoma; Histiocytoma, Malignant Fibrous; Chondrosarcoma; Synovial Sarcoma; Leiomyosarcoma; Liposarcoma; Myosarcoma; Rhabdomyosarcoma; Sarcoma, Alveolar Soft Part; NY-ESO-1; MAGE; MAGE A3; Vaccine; Immunotherapy
MeSH Terms: conditions — Sarcoma; Neoplasms, Connective and Soft Tissue; Fibrosarcoma; Neurofibrosarcoma; Histiocytoma; Histiocytoma, Malignant Fibrous; Chondrosarcoma; Sarcoma, Synovial; Leiomyosarcoma; Liposarcoma; Myosarcoma; Rhabdomyosarcoma; Sarcoma, Alveolar Soft Part | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous dendritic cell vaccine (Experimental): Autologous dendritic cell vaccine loaded with allogeneic tumor lysate expression of cancer testis antigens
  Interventions: Biological: Autologous dendritic cell vaccine

INTERVENTIONS:
Biological: Autologous dendritic cell vaccine — Autologous dendritic cell vaccine loaded with allogeneic tumor lysate expression of cancer testis antigens
  Other Names: Autologous dendritic cell vaccine loaded with allogeneic tumor lysate expression of cancer testis antigens; CTA vaccine; DC vaccine; DC CTA vaccine

SUMMARY:
The purpose of this study is to achieving a six-month progression free survival (PFS) of patients receiving autologous dendritic cell vaccine (ADKV) loaded with allogeneic tumor lysate expression of cancer-testis antigens (CTA) in patients with soft tissue sarcomas

DETAILED DESCRIPTION:
Vaccination is carried out on the planned days ± 3 days

1. All examinations must be performed before the vaccine is administered.

   * Full physical examination.
   * Assessment of vital signs (blood pressure, temperature, heart rate), the general condition of the patient and physical activity.
   * Evaluation of concomitant therapy.
   * Assessment of vital signs.
   * Laboratory safety and immunological indicators
   * Assessment of adverse events, symptoms and syndromes of the disease.
2. Introduction of CV in accordance with the dose determined for a given vaccination (see section 9.2. - procedures for delivery and use)
3. After administration, patients are observed for at least 1 hour. An assessment of vital indicators. Undesirable effects detected at the introduction are recorded.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 or older
* ECOG performance score 0 or 1
* Histologically proven soft tissue sarcoma
* Unresectable or metastatic soft tissue sarcoma
* Ability to give written informed consent
* Objective measured and measurable tumor lesions
* The failure of standard therapy
* Adequate amount of material for genetic research
* No active or chronic infection with HIV, Hepatitis B or Hepatitis C
* Men/Women of childbearing potential must use adequate contraception
* Hematology, liver function and renal function lab tests within required parameters

Exclusion Criteria:

* Untreated or uncontrolled brain metastases.
* History of other active malignancy within last 2 years, except adequately treated other soft tissue sarcoma.
* Autoimmune disease (vitiligo is not a basis for exclusion).
* Serious uncontrolled medical disorder or active infection that would impede treatment.
* Underlying medical or psychiatric condition that would cause administration vaccine
* Any non-oncology vaccine therapy up to 1 month before or after any dose of vaccine
* Concomitant therapy with IL-2, interferon, other non-study immunotherapy, or cytotoxic chemotherapy; immune-suppressive agents within 30 days of registration; other investigational therapies; chronic use of systemic corticosteroids (however, a low stable dose steroid for mild brain edema or adrenal insufficiency is allowed; topical and inhaled standard dose corticosteroids are allowed).
* Dementia or significantly altered mental status that would prohibit understanding or rendering of informed consent and compliance with protocol requirements.
* Pregnant or breastfeeding women.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g. infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-06; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Achieving a six-month progression free survival (PFS) of patients receiving ADKV with soft tissue sarcomas | 6 month
  Achieving a six-month time to progression (PFS) 40% of patients receiving ADKV loaded with allogeneic tumor lysate expressing PTA in patients with soft tissue sarcomas

SECONDARY OUTCOMES:
Median progression-free survival | 6 month
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works
Median overall survival | 6 month
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that half of the patients in a group of patients diagnosed with the disease are still alive. In a clinical trial, measuring the median overall survival is one way to see how well a new treatment works
Objective response rate | 6 mounth
  The percentage of patients whose cancer shrinks or disappears after treatment.
Assess biological response of tumors | 6 mounth
  Сhanging level of T lymphocytes subpopulation in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Komarov, PhD, Study Chair — N. N. Petrov Research Institute of oncology
Locations (1):
- N. N. Petrov Research Institute of oncology, Saint Petersburg, Russia